CLINICAL TRIAL: NCT03526562
Title: Exercise Prescription Dose for Castration Resistance Prostate Cancer Patients: a Phase I Prescription Dose Escalation Trial
Brief Title: Exercise Prescription Dose for Castration Resistance Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2017/1099
Record Dates: First submitted 2018-03-28; First posted 2018-05-16 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Prostatic Neoplasms; Exercise; Castration-resistant Prostate Cancer; Physical Activity
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: phase I study with an exercise prescription as intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm phase I trial with 3 exercise dose-escalation arms (Experimental): exercise dose-escalation: aerobic, resistance and flexibility training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise according to dose escalation

SUMMARY:
Recent drug improvement (e.g. abiraterone or enzalutamide) for castration resistant prostate cancer (CRPC) patients has improved survival. As treatment strategies improve and patients live longer, patients must cope with their treatment-induced adverse effects. Improving levels of physical activity (PA) and less amounts of sitting time (e.g. sedentary behavior, SB) could have a positive impact on patient's health, non-cancer mortality, and quality of life and potentially improve survival.

The role of PA has not yet been examined in CRPC patients, which is a clear unmet need. No specific PA guidelines exist for CRPC patients, but specific guidelines are warranted because of advanced disease stage, reduced performance score and comorbidity. It is to be expected that the PA level of CRPC patients is lower compared to non-CRPC patients receiving androgen deprivation therapy (ADT).

This study aims to determine the optimal starting physical therapy prescription in CRPC patients receiving second line hormone treatment.

DETAILED DESCRIPTION:
CRPC patients receiving second-line hormone treatment at Ghent University Hospital are invited to participate in this phase I 3+3 dose escalation design (escalation to next exercise dose per 3 study patients). The prescription start dose is 15min. aerobic training (50-80% maximum heart rate (HRmax). warm-up and cooling-down and 65-80%HRmax. core), 1 set with 8-10 reps. resistance training (50-60% one repetition maximum (1RM), 8 exercises) and 1 set (30s.) with 2 reps. flexibility training (5 exercises). Factors determining compliance for the dose are tolerance and safety. Tolerance for the exercise prescription will be assessed with the Borg scale of perceived exertion after every exercise. Compliant for tolerance is a score ≤16. Safety will be assessed by the visual analogue scale (VAS) (assessed by the patient) for pain and the CTCAE criteria (assessed by a trained health care provider) for bone pain after every exercise. Compliant for safety is ≤3 VAS for exercise-induced pain and <grade 2 according to the CTCAE criteria.

ELIGIBILITY:
Inclusion Criteria:

* CRPC patients with second-line hormone treatment
* Able to walk 400 meters without help from another person
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (those conditions should be discussed with the patient before registration in the trial)
* ≥4 weeks since any major surgery and fully recovered before patient registration
* Written informed consent must be given according to International conference on harmonization Good Clinical Practice and national regulation.

Exclusion Criteria:

* Musculoskeletal, cardiovascular or neurological comorbidity that prevent the patient to participate in an exercise program
* Painful bone metastases (VAS) at the time of inclusion
* Unstable bone metastases (SINS classification) at time of inclusion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose based on tolerance | change before and after 1 exercise session (at one day)
  Maximum tolerated dose will be assessed by borg scale of perceived exertion.
Maximum tolerated dose based on safety | change before and after 1 exercise session (at one day)
  Maximum tolerated dose will be assessed by CTCAE
Maximum tolerated dose based on safety | change before and after 1 exercise session (at one day)
  Maximum tolerated dose will be assessed by VAS

SECONDARY OUTCOMES:
Functionality | baseline
  Functionality will be assessed by the Karnofsky Performance Status
Pain | baseline
  Pain will be assessed by the Brief pain inventory (BPI) questionnaire
Health Related quality of Life general | baseline
  HRQoL will be assessed by the EORTC quality of life (QLQ) C30 questionnaire
Health Related quality of Life disease specific | baseline
  HRQoL will be assessed by the EORTC quality of life prostate 25 questionnaire
Physical activity level by International Physical Activity Questionnaire (IPAQ) | baseline
  Physical activity level will be assessed by the IPAQ questionnaire
Physical activity level by Godin | baseline
  Physical activity level will be assessed by the Godin Leisure questionnaire
Body composition | baseline
  Body composition will be assessed by 8-point bioelectrical impedance analysis
Physical performance | baseline
  Physical performance will be assessed by the 400m walk test
Physical performance by time up and go | baseline
  Physical performance will be assessed by the time up and go test
Physical performance by 6m walk | baseline
  Physical performance will be assessed by the 6-meter walk test usual and fast pace
Physical performance by 6 m walk backward | baseline
  Physical performance will be assessed by the 6 meter backward walk
Physical performance by Cardiopulmonary Exercise Testing (CPET) | baseline
  Physical performance will be assessed by the CPET
Balance by four square test | baseline
  Balance will be assessed by the four square test
Balance by chair rise test | baseline
  Balance will be assessed by the chair rise test
Motivation 1 | baseline
  Motivation will be assessed by the stages of change theory
Motivation 2 | baseline
  Motivation will be assessed by the Exercise Motivation Inventory questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital ghent, Ghent, Oost-Vlaanderen, Belgium